CLINICAL TRIAL: NCT04705571
Title: Clinical Evaluation of Fractional Bi-Polar Radio-Frequency for Symptoms of Stress Urinary Incontinence and Vulvovaginal Atrophy
Brief Title: Clinical Evaluation of Fractional Bi-Polar RF for Symptoms of SUI and Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO609885A
Record Dates: First submitted 2020-12-24; First posted 2021-01-12 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-01

CONDITIONS: Stress Urinary Incontinence; Vulvovaginal Signs and Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive 1 treatment with the MorpheusV Applicator according to the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MorpheusV Applicator (active) (Experimental)
  Interventions: Device: MorpheusV Applicator

INTERVENTIONS:
Device: MorpheusV Applicator — 1 treatment with the MorpheusV Applicator

SUMMARY:
Clinical Evaluation of Fractional Bi-Polar Radio-Frequency for Symptoms of Stress Urinary Incontinence and Vulvovaginal Atrophy

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the safety and efficacy of the MorpheusV Applicator for Symptoms of Stress Urinary Incontinence and Vulvovaginal Atrophy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.

  * Female subjects, 35 and 75 years of age at the time of enrolment with primary and moderate to severe symptoms of SUI, who had scored at least 6 out of 12 according to severity index developed by Sandvik
  * She has produced a leak during the bladder "cough" stress test.
  * 18 out of 27 for the Stress Incontinence Questions and were confirmed as having predominant SUI on the Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire completed at the screening assessment.
  * General good health confirmed by medical history and skin examination of the treated area.
  * The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* - Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance, unless deep enough in the periostal plane.
* Current or history of cancer, or premalignant condition in the treatment area.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Simultaneous participation in another investigator drug or device study or completion of the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
* Six months delay is required if other recent treatments like light, CO2 laser or RF were performed on the same area.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
An objective change as measured by standardized cough stress test | Day 0, Month 6
  An objective change as measured by standardized cough stress test performed in standing position before treatment and at 6 months (6M FU) after the treatment
An objective evaluation of vaginal atrophy/estrogenization | Day 0, month 6
  An objective evaluation of vaginal atrophy/estrogenization measured by the globally validated "Vaginal Health Index" (VHI) score at 6M FU compared to Baseline.
The effect of the treatment on urinary symptoms and quality of life by means of the Incontinence Quality of Life (IQOL) Questionnaire | Day 0, month 6
  The effect of the treatment on urinary symptoms and quality of life by means of the Incontinence Quality of Life (IQOL) Questionnaire. Administered at baseline and at 6M FU.
The effect of the treatment on urinary symptoms by means of Urogenital Distress Inventory 6 Questionnaire | day 0, month 6
  The effect of the treatment on urinary symptoms by means of Urogenital Distress Inventory 6 Questionnaire. Administered at baseline and at 6M FU.
The effect of the treatment on urinary symptoms by means of Bladder voiding diary after the treatment | Day 0, month 6
  The effect of the treatment on urinary symptoms by means of Bladder voiding diary after the treatment, and at 6M FU versus baseline.
The effect of the treatment on urinary symptoms by means of Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire | Day 0, month 6
  The effect of the treatment on urinary symptoms by means of Medical, Epidemiologic, and Social Aspects of Aging Urinary Incontinence (MESA) Questionnaire at 6M FU versus baseline.
Evaluation of histological changes to vaginal canal tissue | Day 0, month 3
  Evaluation of histological changes to vaginal canal tissue taken immediately post treatment and at 3M FU versus baseline. (for 5 subjects)

SECONDARY OUTCOMES:
Occurrence of expected post treatment immediate response | day 0, through study completion, on average 6 months
  Occurrence of expected post treatment immediate response including erythema and edema and during all study period based on predefined scale
Discomfort scale | day 0
  A 10cm visual analog scale from 0 (no discomfort) to 10 (worst possible discomfort) to measure discomfort associated with probe insertion, and RF energy application
Adverse Events | Through study completion, an average of 6 months
  Number, severity and type of any adverse event recorded throughout the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Blusewicz, MD, Principal Investigator — Advanced Women's Care of the Lowcountry, PC
Locations (2):
- United States (2):
  - Miklos and Moore Urogynecology, Alpharetta, Georgia
  - Advanced Women's Care of the Lowcountry, PC, Bluffton, South Carolina

IPD SHARING:
Plan to Share IPD: No